CLINICAL TRIAL: NCT01815385
Title: Early Life Exposure to Polycyclic Aromatic Hydrocarbons: Metabolic Perturbations and Epigenetic Biomarkers
Brief Title: Epigenetic and Developmental Effects of In Utero Exposure to Environmental Toxicants
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Mamta Fuloria, Associate Professor, Pediatrics, Montefiore Medical Center
Other Study IDs: 12-12-428; 1-13-CE-06 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Full Term Infants; Environmental Exposures; Adiposity
Keywords: Term gestation; Environmental exposure; Benzo(a)pyrene; Polycyclic aromatic hydrocarbons; Adiposity; Cytosine methylation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood sample Cord blood sample Infant saliva Peripheral blood sample from enrolled patients at 12 and 24 months of age
Oversight: Data Monitoring Committee: No

SUMMARY:
Metabolic diseases such as obesity and diabetes are modern day epidemics. Early life exposure to an adverse developmental environment, including environmental toxins, are linked to increased susceptibility to obesity, metabolic syndrome and type 2 diabetes. Although the mechanisms underlying the fetal origins of metabolic disease are poorly understood, strong evidence suggests that alterations in the epigenome play a critical role in this process. The central hypothesis of this proposal is that intrauterine exposure to benzo[a]pyrene leads to epigenetic changes which will have functional consequences and may be a marker for, or may contribute to, increased susceptibility to adverse outcomes in childhood including increased adiposity and the subsequent development of obesity, metabolic syndrome or diabetes. The goals of this proposal are to: 1) determine benzo[a]pyrene levels in umbilical cord blood of newborns, 2) determine whether benzo[a]pyrene exposure during pregnancy correlates with early onset of obesity and metabolic disease by examining the children at 12 and 24 months of age, 3) determine whether in utero benzo[a]pyrene exposure programs metabolic disease through alterations in DNA methylation and gene expression, and 4) determine the plasticity of the DNA methylation patterns in the same offspring at 12 months of age. The long-term goal of this project is to define biomarkers that identify neonates at "high-risk" for diminished attainment of full health potential, who can then be targeted for preventative measures.

ELIGIBILITY:
Inclusion Criteria:

* Infants whose mothers were followed by the Obstetric Department at MMC, and
* Deliver a single healthy live term infant

Exclusion Criteria:

* Multiple gestation,
* Maternal depression,
* History of maternal smoking in the 3rd trimester of pregnancy,
* Infants in extremis,
* Apgar score <7 at 5 min and umbilical artery pH ≤7.25,
* Chromosomal/congenital abnormalities,
* Congenital infections, and
* Inborn errors of metabolism

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother-baby pairs will be recruited.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Measure indices of adiposity in enrolled patients | up to 24 months
  Assessments will be performed within 72 hours of birth and at 1 and 2 years of age.
Measure benzo(a)pyrene levels in blood samples | up to 12 months of age
  Benzo(a)pyrene levels will be measured in cord blood samples obtained at birth and in peripheral blood samples obtained at 12 months of age.
Measure tobacco by-products in blood samples | up to 12 months of age
  Levels of tobacco by-products will be measured in cord blood samples obtained at birth and in peripheral blood samples obtained at 12 months of age.
Characterize cytosine methylation changes in CD3+ T-lymphocytes | up to 12 months of age
  Cytosine methylation changes in CD3+ T-lymphocytes will be characterized in cord blood and in a peripheral blood sample obtained at 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Fuloria, MD, Principal Investigator — Montefiore Medical Center; Maureen Charron, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center - Jack D. Weiler Division, The Bronx, New York, United States